CLINICAL TRIAL: NCT05193877
Title: Autologous Bone Marrow Aspirate Concentrate Injection for the Treatment of Early Osteoarthritis: a Randomized Controlled Trial, Ibn-Sina Hospital, Baghdad 2022
Brief Title: Autologous Bone Marrow Aspirate Concentrate Injection for the Treatment of Early Osteoarthritis:Baghdad 2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Global Stem Cell Center, Baghdad (Industry)
Responsible Party: Principal Investigator, abdulmajeed hammadi, global stem cell center baghdad, Global Stem Cell Center, Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ibn-sina protocol
Record Dates: First submitted 2021-12-24; First posted 2022-01-18 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Treatment Complication

STUDY DESIGN:
Intervention Model Description: double blind
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment with autologous bone marrow aspirate concentrate (Active Comparator): autologous bone marrow aspirate is taken under local anesthesia to be centrifuged and the concentrate given intra articularly in knee joint
  Interventions: Procedure: autologous bone marrow aspirate concentrate by centrifugation
- control (Sham Comparator): control group given analgesics only
  Interventions: Procedure: autologous bone marrow aspirate concentrate by centrifugation

INTERVENTIONS:
Procedure: autologous bone marrow aspirate concentrate by centrifugation — 50 cc bone marrow aspirates concentrate after centrifugation with final volume up to 7 cc.
  Assess total nucleated count and viability. Bone marrow aspirate concentrate is chosen as a source of mesenchymal stem cells, because of safe and easy procedure.
  Bone marrow aspiration is done under local or general anesthesia, depending on the individual case. Around 50 cc of bone marrow is aspirated from the posterior iliac crest after proper sterilization using bone marrow aspiration needle (size according to the patient) and collected in heparinized syringes. Mononuclear cells (MNCs) are obtained by centrifugation. The isolated MNCs are checked for viability manually and confirmed on automated cell count machine.
  The separated MNCs is administered intra-articularly immediately after centrifugation.

SUMMARY:
We present a randomized controlled trial (RCT) to assess the efﬁcacy of autologous bone marrow aspirate concentrate BMAC of 1.8x 10 9 median cellular content in the treatment of early symptomatic knee OA. We use 2 injections 2 months apart (8).

DETAILED DESCRIPTION:
1. To evaluate the efficacy of bone marrow aspirate concentrate (BMAC) therapy on pain, function and disease modification in knee osteoarthritis.
2. To determine the potential of BMAC therapy to achieve disease modification, as detected through radiological examination using magnetic resonance imaging (MRI) techniques.
3. Methodology:

A randomized controlled trial will be held in Ibn-Sina training hospital in Baghdad. All participants will complete written informed consent. The study will be a single centered trial.

The trial design will consist of 60 participant randomly and equally allocated to control and treatment group by simple random sampling. Participants will not be blinded to their treatment allocation. Control group will receive conventional treatment only. Intervention group will receive (2 injections) intra-articular injections of (4cc) per joint at (8 weeks' interval).

Intervention:

50 cc bone marrow aspirates concentrate after centrifugation with final volume up to 7 cc.

Assess total nucleated count and viability. Bone marrow aspirate concentrate is chosen as a source of mesenchymal stem cells, because of safe and easy procedure.

Bone marrow aspiration is done under local or general anesthesia, depending on the individual case. Around 50 cc of bone marrow is aspirated from the posterior iliac crest after proper sterilization using bone marrow aspiration needle (size according to the patient) and collected in heparinized syringes. Mononuclear cells (MNCs) are obtained by centrifugation. The isolated MNCs are checked for viability manually and confirmed on automated cell count machine.

The separated MNCs is administered intra-articularly immediately after centrifugation.

Place:

Bone marrow aspiration and centrifugation procedure is done in clean area, in operation room HEPA filtered with all instruments included. Cell count viability and flow cytometry can be sent to nearby lab.CD markers (90, 44,29,105,34).

Instruments:

Bone marrow aspiration kit, centrifuge, automated cell counter.

Sample size and sampling technique:

The conventional treatment is usually classic treatment .

Statistical analysis:

Raw data will be summarized, and presented in appropriate table. The statistical analysis will be carried out using SPSS (statistical package for social science) software version 25

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of Osteoarthritis according to Kellgren and Lawrence Criteria stage II-III.

  * Radiological grading of osteoarthritis of the knee determined by qualified radiologist using MOAKS scoring system.
  * Primary osteoarthritis not responsive to conventional treatment and physiotherapy.
  * A minimum pain score of 5 on an 11-point numerical scale.
  * Age >55 years

Exclusion Criteria:

* Pregnancy and breast feeding.
* Knee symptom due to other condition like tumor or referred pain from lumbar spine.
* MRI confirmed displaced meniscal tear
* MRI confirmed Grade IV chondral loss.
* Previous knee surgery within the last 12 months.
* Previous intra-articular injectable therapies within the last 6 months
* History of severe systemic illness.
* Active neoplasm under treatment in the last 12 months- Health conditions including known allergy to local
* Bleeding tendency.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
clinical | 6 months
  improvement in pain scale WOMAC

SECONDARY OUTCOMES:
radiological proof | 6 months-1 year
  MRI of the knee joint to monitor effect

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No